CLINICAL TRIAL: NCT05752175
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of WPV01 in Patients With Mild/Moderate COVID-19 Infection
Brief Title: Study of WPV01 Compared With Placebo in Patients With Mild/Moderate COVID-19 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Westlake Pharmaceuticals (Hangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WPV01-CP-02
Record Dates: First submitted 2023-03-01; First posted 2023-03-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WPV01 (Experimental)
  Interventions: Drug: WPV01
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WPV01 — WPV01 tablets
  Arms: WPV01
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of WPV01 in patients with mild/moderate COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years of age when signing ICF;
2. Initial onset at least 1 of 11 COVID-19 symptoms within 48 hours before randomization;
3. Within three days before randomization, the RT-PCR test of specimens such as nasal and pharyngeal swabs must be positive for SARS-CoV-2 or the rapid antigen test must be positive, and also the patiets should meet the diagnostic criteria for mild or moderate cases as defined in the Diagnosis and Treatment Protocol for COVID-19 (Trial Version 10) issued by the National Health Commission of China;
4. Fertile participants must agree to take effective contraceptive measures;
5. Participants who understand and agree to comply with planned study procedures，voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Known allergy to any ingredient in the study treatment drug;
2. Patients who meet the diagnostic criteria for severe or critical cases of COVID-19 as defined in the Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 10) issued by the National Health Commission of China at the time of randomization;
3. Obvious abnormal liver function (ALT or AST ≥ 3ULN, or total bilirubin ≥1.5ULN);
4. On dialysis or combined with moderate to severe kidney injury;
5. Patients with compromised immune system;
6. Patients with acute exacerbation of chronic respiratory disease at screening, including bronchial asthma, chronic obstructive pulmonary disease;
7. Patients with suspected or confirmed concurrent active systemic infection other than COVID-19 at screening;
8. Any comorbidity requiring surgery within 14 days prior to study entry, or that is considered life threatening within 30 days prior to study entry, as determined by the investigator;
9. Has received or is expected to receive COVID-19 monoclonal antibody or convalescent COVID-19 plasma during study treatment;
10. Has received treatment with antivirals against SARS-CoV-2 within 14 days prior to randomization;
11. Has received any novel coronavirus infection vaccine within 1 week prior to randomization;
12. Current or expected use of strong CYP3A4 inducers, inhibitors or medications that are highly dependent on CYP3A4 for clearance;
13. Difficulty swallowing or a history of gastrointestinal disorders that severely interfere with drug absorption;
14. BMI≥30 kg/m2;
15. Pregnant, lactating women or those with a positive pregnancy test;
16. Previous administration with any investigational drug within 3 months before the study drug administration;
17. Patients who are judged by the investigator to be unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Changes in viral load | Baseline through Day 7
  Change of viral load compared to the baseline

SECONDARY OUTCOMES:
Change in the total score of COVID-19 symptoms | Baseline through Day 14
  Change in the total score of COVID-19 symptoms compared to the baseline
Change in the score of each COVID-19 symptom | Baseline through Day 14
  Change in the score of each COVID-19 symptom compared to the baseline
Change of EuroQol Questionnaire - 5 Dimension (EQ-5D) | Baseline through Day 14
  Change of EuroQol Questionnaire - 5 Dimension (EQ-5D) compared to the baseline
percentage of patients who reached the sustained clinical recovery of COVID-19 symptoms in every visit | Baseline through Day 14
  percentage of patients who reached COVID-19 symptoms scores of 0 for two consecutive days in every visit
Time to the first negative SARS CoV-2 test result | Baseline through Day 14
  The time from the start of treatment to the time when the first negative SARS CoV-2 qPCR result showed CT value ≥35
progression of COVID-19 infection | Baseline through Day 14
  the percentage of patients who progressed to severe/critical COVID-19 or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Hainv Gao, Principal Investigator — Shulan (Hangzhou) Hospital
Locations (1):
- Shulan(Hangzhou) Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided
6 months after summary data has been published, sponsor will share the IPD and additional supporting information after internal approval process.